CLINICAL TRIAL: NCT03947827
Title: Minocycline As Adjunctive Treatment for Treatment Resistant Depression: a Double Blind, Placebo-controlled, Randomized Trial
Brief Title: Minocycline As Adjunctive Treatment for Treatment Resistant Depression
Acronym: MINDEP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Ishrat Husain, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 135/2018
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Minocycline; Neuroinflammation; Microglial Activation; Biomarker
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; cyclopia sequence; Neuroinflammatory Diseases | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, their families, referring clinicians, lab workers and research assistants carrying out assessments will be concealed from allocation. Once randomized, pharmacy at the Centre for Addiction and Mental Health (CAMH) will be informed by email and deliver medication to the patient. An independent study psychiatrist will manage any clinical concerns and will be blind to treatment allocation. To assess the integrity of blinding procedures, participants and independent raters will be asked to complete a conventional guess form asking whether they believe participants received Minocycline or placebo as a treatment after the final ratings have been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Minocycline will start at an oral dose of 100mg daily and will be increased after one week to 100mg twice daily.
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Placebo capsules will start at one capsule daily, and will be increased after one week to one capsule twice daily
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Participants will be randomized to receive either Minocycline or placebo added to standard oral antidepressants.
  Other Names: Apo-Minocycline

SUMMARY:
Major depressive disorder (MDD) is a leading cause of disability worldwide. Up to 50% of patients experience treatment resistant depression (TRD), which accounts for a vast majority of disease burden. Current medications for TRD have limited efficacy and can be associated with intolerable side effects. Therefore, there is a need for finding new treatment targets. Accumulating evidence suggests some patients with MDD including those with TRD, display brain inflammation. Thus, patients with TRD may benefit from medications that can reduce this inflammation. Minocycline is an antibiotic which can cross the blood-brain barrier and has effects on several systems implicated in depression. The principal investigator led the first pilot study of minocycline as an add-on treatment in TRD demonstrating that it led to a significant reduction in depressive symptoms compared to placebo and these findings require replication in a larger sample to confirm the efficacy and tolerability of this treatment approach.

This study is a 12 week, double-blind, placebo-controlled trial of minocycline as add-on treatment for patients suffering from a major depressive episode who have failed to respond to antidepressant treatment, confirmed by the Structured Clinical Interview for DSM-5 (SCID-5) and the Antidepressant Treatment History Form (ATHF) at screening. After screening and randomization to the two parallel arms of the trial, 50 patients will receive minocycline added to treatment as usual (TAU) and 50 patients will receive placebo added to TAU. Clinical assessment will include the Hamilton Depression Rating Scale (HRSD-17), Clinical Global Impression scale (CGI), World Health Organization Quality of Life Short Form (WHOQOL-BREF), and Generalized Anxiety Disorder scale (GAD-7), administered at each study visit (baseline, week 2, 6, and 12). Side effects checklists will be undertaken at each visit. Minocycline will be started at 100 mg once daily and will be increased to 100 mg twice daily at two weeks. Secondary outcomes include inflammatory biomarkers measured at baseline, weeks 6 and 12.

This trial will provide further evidence of minocycline's efficacy and acceptability as a treatment option for patients with TRD and provide insights into its mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Voluntary and competent to consent to treatment
3. DSM-5 diagnosis of non-psychotic MDD, single or recurrent, based on the SCID-5
4. Male or female aged between 18-80
5. Total score > 3 on ATHF
6. Baseline HRSD-17 score > 14
7. Able to adhere to study schedule
8. If female of childbearing potential, currently on a medically acceptable form of birth control (oral contraceptives, contraceptive injections, IUD, contraceptive patch, male partner sterilization, abstinence, or barrier methods plus spermicide)
9. Currently taking one of the following standard antidepressants: Escitalopram, Citalopram, Sertraline, Venlafaxine, Duloxetine, Mirtazapine or Bupropion
10. Been on same dose of all psychotropic medications for > 4 weeks prior to enrolment

Exclusion Criteria:

1. DSM-5 substance use disorder within past 3 months, moderate or severe, based on SCID-5
2. Concomitant major unstable medical illness
3. Pregnancy or intent to become pregnant during study period
4. DSM-5 diagnosis of psychotic disorder, bipolar disorder, obsessive-compulsive disorder (OCD), post-traumatic stress disorder (PTSD) within last year
5. DSM-5 diagnosis of borderline personality disorder (BPD)
6. Possible or probable dementia
7. Prior or current intolerance or contraindication to tetracyclines
8. Abnormal readings in hematology, liver, or renal function tests
9. Have Myasthenia Gravis
10. Concomitant treatment with anticoagulants, diuretics, retinoids, ergot alkaloids, antacids containing aluminium/calcium/magnesium, bismuth and zinc salts, or quinapril

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 12 weeks
  Changes from baseline to week 12 on the 17-item Hamilton Rating Scale for Depression (HRSD-17).

SECONDARY OUTCOMES:
Response rate | 12 weeks
  Reduction of 50% or more in HRSD score from baseline to week 12
Remission rate | 12 weeks
  Final HRSD score < 8
Anxiety symptoms | 12 weeks
  Changes from baseline to week 12 in Generalized Anxiety Disorder scale (GAD-7)
Self-reported perception of quality of life | 12 weeks
  Changes from baseline to week 12 in World Health Organization Quality of Life Short Version (WHOQOL-BREF)
Clinician-rated illness severity | 12 weeks
  Changes from baseline to week 12 in Clinical Global Impression scale (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Ishrat Husain, MBBS, MD(Res.), Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Husain MI, Cullen C, Umer M, Carvalho AF, Kloiber S, Meyer JH, Ortiz A, Knyahnytska Y, Husain MO, Giddens J, Diniz BS, Wang W, Young AH, Mulsant BH, Daskalakis ZJ. Minocycline as adjunctive treatment for treatment-resistant depression: study protocol for a double blind, placebo-controlled, randomized trial (MINDEP2). BMC Psychiatry. 2020 Apr 15;20(1):173. doi: 10.1186/s12888-020-02553-9. PMID 32295565